CLINICAL TRIAL: NCT05863260
Title: Tislelizumab (Anti-PD-1) Combined With Definitive Chemoradiotherapy in Recurrent Cervical Cancer (PILOT-2020-511): a Single-arm, Phase 2 Trial
Brief Title: Tislelizumab Combing Chemoradiotherapy in Recurrent Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Professor, Fudan University
Other Study IDs: PILOT-2020-511
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cervical Cancer; Immune Checkpoint Inhibitor; Chemoradiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Paclitaxel 135mg / m2d1 + cisplatin 60mg / m2d1 (cisplatin resistance or cisplatin intolerance changed to carboplatin AUC = 5d1), q3w × 4 and Standard IMRT and radiotherapyTislelizumab 200mg, IV, q3w, the day before radiotherapy
  Interventions: Drug: Treatment Group

INTERVENTIONS:
Drug: Treatment Group — Treatment Group

SUMMARY:
Tislelizumab combined with chemoradiotherapy in the treatment of recurrent/ metastasis cervical cancer: a single arm,single center， phase ii and observational clinical study

DETAILED DESCRIPTION:
Tislelizumab combined with chemoradiotherapy in the treatment of recurrent/ metastasis cervical cancer: a single arm,single center， phase ii and observational clinical study

ELIGIBILITY:
Inclusion Criteria:

1. For patients with recurrent or metastatic cervical cancer after initial standard treatment (including radical surgery or radical radiotherapy), the lesions are located out of the field of previous radiotherapy, with no more than 5 recurrent or metastatic foci, and the radiotherapy is feasible according to the evaluation of radiotherapy physician; and at least 1 lesion (without previous radiotherapy) meets the target lesion standard of RECIST 1.1;
2. Cervical adenocarcinoma, squamous cell carcinoma or adenosquamous cell carcinoma confirmed by previous histology;
3. Surgical resection is not recommended for recurrent lesions, or patients choose not to accept surgery voluntarily;
4. The researchers evaluated the suitability of radiotherapy
5. ECoG 0-1; life expectancy > 6 months;
6. Aged 18-70 years;
7. No serious allergic history;
8. Hemoglobin > 100 g / L, WBC > 3.5 * 10 ^ 9 / L, neutrophils > 1.5 * 10 ^ 9 / L, platelets > 100 * 10 ^ 9 / L, Cr < 1.5 * normal upper limit, TB < 2.5 * normal upper limit, AST and Al < 2.5 * normal upper limit, AKP < 2.5 * normal upper limit;
9. Ability to sign informed consent.

Exclusion Criteria:

1. Histologically, small cell (neuroendocrine) cervical cancer, mucinous adenocarcinoma, carcinosarcoma and other pathological types were confirmed;
2. Primary malignant tumor with activity in other parts, except for the following:

   Those who have been cured have no known active disease at least 5 years before the first IP administration, and the potential risk of recurrence is low;

   Fully treat non melanoma skin cancer or malignant nevus without disease signs;

   Fully treated carcinoma in situ, no signs of disease.
3. The recurrent lesions have received chemotherapy, radiotherapy or other anti-tumor treatment;
4. Bone metastasis;
5. Brain metastasis;
6. Pregnant or lactating patients;
7. In the past, there was abnormal thyroid function, and under the condition of drug treatment, thyroid function could not be maintained in the normal range;
8. Diagnosis of immune deficiency or treatment with chronic systemic steroids (doses more than 10 mg per day of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before enrollment;
9. Patients with active autoimmune diseases need systemic treatment in the past 2 years;
10. A history of (noninfectious) pneumonia requiring steroids or current pneumonia;
11. There are active infections that need systematic treatment;
12. Known history of human immunodeficiency virus (HIV) infection;
13. Known history of hepatitis B or known active hepatitis C virus infection;
14. Known history of active tuberculosis (TB);
15. Uncontrolled comorbidities, including but not limited to: persistent or active infection, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled diabetes, uncontrolled arrhythmias, active interstitial lung disease (ILD), severe chronic gastrointestinal disease with diarrhea, or may limit compliance with study requirements, leading to AE Mental / social problems that significantly increase or affect the ability of subjects to provide written informed consent;
16. 14 days before admission, the operation was too large and had not recovered;
17. Participate in other clinical trials at present or within 28 days before selection;
18. Any indications, including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1 and anti-PD-L2 antibodies or therapeutic anti-cancer vaccines, were treated by immunomediated therapy prior to the study;
19. Any synchronous chemotherapy, research drug, biological product, or hormone therapy used to treat tumors. Hormone therapy can also be used to treat non tumor related diseases (e.g., hormone replacement therapy);
20. Allogeneic tissue / solid organ transplantation was carried out.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with recurrent or metastatic cervical cancer after initial standard treatment (including radical surgery or radical radiotherapy), the lesions are located out of the field of previous radiotherapy, with no more than 5 recurrent or metastatic foci, and the radiotherapy is feasible according to the evaluation of radiotherapy physician; and at least 1 lesion (without previous radiotherapy) meets the target lesion standard of RECIST 1.1
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Objective response rate

SECONDARY OUTCOMES:
1-year PFS | 1 year
  1-year PFS
1-year OS | 1 year
  1-year OS

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China